CLINICAL TRIAL: NCT00755976
Title: Phase II Trial of the Multi-Drug Resistance Protein Modulating Agent Sulindac in Combination With Epirubicin in Patients With Advanced Melanoma
Brief Title: Sulindac and Epirubicin in Treating Patients With Metastatic Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-03 ICORG; ICORG-06-03; EUDRACT-2006-006051-12; EU-20876; NCT00632177 (obsolete NCT alias)
Record Dates: First submitted 2008-09-13; First posted 2008-09-19 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2012-10

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Epirubicin; Sulindac; Immunologic Techniques

ARMS (1):
- Epirubicin hydrochloride (75mg/m2 i.v.) Sulindac: 600mg (Experimental)
  Interventions: Drug: epirubicin hydrochloride; Drug: sulindac; Other: immunologic technique

INTERVENTIONS:
Drug: epirubicin hydrochloride
Drug: sulindac
Other: immunologic technique

SUMMARY:
RATIONALE: Sulindac may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as epirubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sulindac together with epirubicin may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving sulindac together with epirubicin works in treating patients with metastatic malignant melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the non-comparative efficacy of sulindac and epirubicin hydrochloride in patients with metastatic malignant melanoma.

Secondary

* To characterize the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral sulindac 2 hours prior to receiving epirubicin hydrochloride IV over 15 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Previously collected tumor blocks are assessed for cancer resistance markers by IHC.

After completion of study treatment, patients are followed for 1 month, and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant melanoma

  * Metastatic disease
* Tumor block available for resistance marker analysis
* Measurable or evaluable disease
* No active brain metastases except for patients who have undergone successful complete excision of solitary brain metastasis

PATIENT CHARACTERISTICS:

* Karnofsky performance status 80-100%
* ANC > 1 x 10^9/L
* Platelet count > 100 x 10^9/L
* Hemoglobin > 9 g/dL
* Serum bilirubin normal (except in patients with benign congenital hyperbilirubinemia)
* Not pregnant or nursing
* Negative pregnancy test
* Normal cardiac ejection fraction, cardiac wall motion, and ECG
* No active heart disease, including any of the following:

  * Myocardial infarction within the past year
  * Pericarditis
  * Existing hypertension requiring treatment
* No other active serious medical or psychiatric disease
* No prior or concurrent malignancy, other than basal cell carcinoma of the skin , or carcinoma in-situ of the cervix

PRIOR CONCURRENT THERAPY:

* No prior anthracycline or anthracenedione-containing chemotherapy regimen
* No prior cardiac radiotherapy
* No major surgery within the past 2 weeks
* No participation in any clinical trial within the past 4 weeks
* No other concurrent anticancer therapies

  * Concurrent bisphosphonates allowed in patients with bony metastases with extra-osseous measurable or evaluable lesions
* No other concurrent experimental medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To estimate the non-comparative efficacy of this treatment combination in patients with malignant melanoma. Response will be assessed using the RECIST Criteria | Ongoing throughout trial
  The interim analysis will study the objective response to treatment in the first cohort of 29 patients. Response will be assessed according to NCI -Response Evaluation Criteria in Solid Tumors (RECIST) guidelines

SECONDARY OUTCOMES:
Toxicity according to NCI CTCAE v.3.0 | Ongoing throughout trial

CONTACTS AND LOCATIONS:
Overall Officials: John Crown, MD, Principal Investigator — St Vincent's University Hospital, Ireland
Locations (10):
- Ireland (10):
  - Cork University Hospital, Cork
  - Adelaide and Meath Hospital, Dublin Incorporating the National Children's Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St. James's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - National Institute for Cellular Biotechnology at Dublin City University, Dublin
  - Galway University Hospital, Galway
  - Mid-Western Cancer Centre at Mid-Western Regional Hospital, Limerick
  - Waterford Regional Hospital, Waterford